CLINICAL TRIAL: NCT06366672
Title: Evaluating the Durability of the Human Immune Response to the JYNNEOS Modified Vaccinia Ankara-Bavarian Nordic (MVA-BN) Vaccine
Brief Title: Evaluating the Human Immune Response to the JYNNEOS Vaccine
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Philip Mudd, Assistant Professor, Washington University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 202312043
Record Dates: First submitted 2024-04-04; First posted 2024-04-16 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Vaccinia; Virus Diseases
Keywords: T cell; neutralizing antibody; mucosal immunity
MeSH Terms: conditions — Vaccinia; Virus Diseases | interventions — smallpox and monkeypox vaccine modified vaccinia ankara-bavarian nordic; Smallpox Vaccine; Suspensions; Injections, Subcutaneous; Phlebotomy

STUDY DESIGN:
Intervention Model Description: Participants will be vaccinated with MVA-BN according to the FDA-approved labeling and immune responses in the blood, lung mucosa, skin, and bone marrow will be monitored prior to and following vaccination using phlebotomy, research bronchoscopy, skin punch biopsy, and bone marrow aspiration procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- MVA-BN vaccinated (Experimental): MVA-BN vaccine administered: day 0 and day 28 Phlebotomy: within 30 days prior to first vaccine dose, day 0, day 14, day 28, day 35, day 42, day 56, day 90, day 110, day 150, day 210, day 395 Research bronchoscopy: within 30 days prior to first vaccine dose, day 42, day 210, day 395 Skin punch biopsy: within 30 days prior to first vaccine dose, day 42, day 210, day 395 Bone marrow aspiration: within 30 days prior to first vaccine dose, day 56, day 110, day 210, day 395
  Interventions: Biological: JYNNEOS (Smallpox and Monkeypox Vaccine, Live, Nonreplicating) suspension for subcutaneous injection; Procedure: Phlebotomy; Procedure: Research bronchoscopy; Procedure: Skin punch biopsy; Procedure: Bone marrow aspiration

INTERVENTIONS:
Biological: JYNNEOS (Smallpox and Monkeypox Vaccine, Live, Nonreplicating) suspension for subcutaneous injection — live, nonreplicating vaccine delivered according to the FDA approved package insert
Procedure: Phlebotomy — Research blood draw
Procedure: Research bronchoscopy — Outpatient research bronchoscopy with bronchoalveolar lavage and endobronchial biopsy performed with conscious sedation.
Procedure: Skin punch biopsy — Skin punch biopsy performed with topical anesthesia.
Procedure: Bone marrow aspiration — Bone marrow aspiration performed with local anesthesia.

SUMMARY:
This study is designed to evaluate the magnitude and duration of the human adaptive immune response to the JYNNEOS Modified Vaccinia Ankara-Bavarian Nordic (MVA-BN) vaccine in the blood, lung mucosa, skin and bone marrow.

DETAILED DESCRIPTION:
Orthopoxvirus vaccination leads to very high magnitude antigen-specific T cell responses and neutralizing antibody responses that can be detected in blood decades after vaccination. Despite a large number of previous studies of human immune responses to Modified Vaccinia Ankara (MVA) vaccination in blood, very few of these previous studies evaluate the human mucosal immune response to MVA in the lung and skin, or the immune response to MVA vaccination in the bone marrow. The development of methods to explore human immune responses in these key immunologic compartments now allows the evaluation of the induction of immune responses in these human tissues using the MVA vaccine system.

ELIGIBILITY:
Inclusion Criteria:

* 18-60 year old otherwise healthy participants

Exclusion Criteria:

* Prisoners
* Participants unable to provide full written informed consent
* Previous receipt of a smallpox or monkeypox vaccine
* Previous infection with monkeypox
* Receipt of any vaccine in the 28 days prior to the first study procedure or planned receipt of any vaccine outside of those provided in the current study before completion of the study day 42 visit.
* Immunocompromise (primary or secondary due to other medical conditions or medications)
* Previous organ transplant
* Active malignancy
* Pregnancy
* < 4 weeks post-partum or actively breastfeeding
* Female participants who are not actively on hormonal contraception or do not have an intrauterine device in place
* Body Mass Index > 40
* Current smokers
* History of a known chronic pulmonary, cardiovascular, renal, hepatic, hematologic or metabolic disorder. Participants with isolated treated hypertension as the only cardiovascular disorder may be included in the study.
* History of a chronic neurologic or neurodevelopmental condition. This does not exclude potential participants with chronic back pain or previous disk herniation/back surgery, only participants with documented weakness, quadriplegia or paraplegia. This exclusion criterion also does not exclude from the study participants with recurrent migraine headaches as the only chronic neurologic condition.
* Pulse oxygen saturation value of 92% or less on room air at study enrollment or on the day of bronchoscopy
* Any significant infiltrate or pleural effusion on upright posterior-anterior and lateral chest x-ray imaging performed on the day of bronchoscopy
* International Normalized Ratio value greater than 1.4 or a Partial Thromboplastin Time value of greater than 40 seconds at study enrollment
* Platelet count of less than 100,000 at study enrollment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-06-10 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in magnitude of the MVA-BN antigen-specific T cell response in the blood | Change from day 42 to day 395
Change in magnitude of the MVA-BN antigen-specific antibody response in blood plasma | Change from day 42 to day 395

SECONDARY OUTCOMES:
Change in magnitude of the MVA-BN antigen-specific T cell response in the lower airways | Change from day 42 to day 395
Change in magnitude of the MVA-BN antigen-specific antibody response in bronchoalveolar lavage fluid | Change from day 42 to day 395

OTHER OUTCOMES:
Evaluate the magnitude and surface phenotype of T cells in the blood, airspace, and skin over time | Through study completion on day 395
Evaluate the magnitude and surface phenotype of B cells in the blood and bone marrow over time. | Through study completion on day 395

CONTACTS AND LOCATIONS:
Overall Officials: Philip Mudd, MD, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in Saint Louis School of Medicine Emergency Care and Research Core, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No